CLINICAL TRIAL: NCT06345066
Title: A Multiple Dose Combination Study to Evaluate the Safety and Tolerability of Tirzepatide and LY3841136 in Overweight and Obese Participants
Brief Title: A Study of LY3841136 in Overweight and Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18834; J3R-MC-YDAC (Other: Eli Lilly And Company)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Overweight
Keywords: Safety; Tolerability; Body weight
MeSH Terms: conditions — Obesity; Overweight; Body Weight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3841136 + Tirzepatide (Experimental): LY3841136 administered subcutaneously (SC) in combination with tirzepatide given SC.
  Interventions: Drug: Tirzepatide; Drug: LY3841136
- Placebo + Tirzepatide (Placebo Comparator): Placebo administered SC in combination with tirzepatide given SC.
  Interventions: Drug: Tirzepatide; Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC.
Drug: LY3841136 — Administered SC.
  Arms: LY3841136 + Tirzepatide
Drug: Placebo — Administered SC.
  Arms: Placebo + Tirzepatide

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of LY3841136 when administered in combination with tirzepatide in overweight and obese patients. The study will last up to approximately 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation
* Have a stable body weight and Body Mass Index in range of 27 to 45 kilogram per meter square (kg/m²).
* Have clinical laboratory test results within normal reference range
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have type 1 or type 2 diabetes mellitus
* Have an abnormal 12-lead electrocardiogram (ECG)
* Have a history or presence of psychiatric disorders
* Have abnormal blood pressure and pulse rate
* Are currently enrolled in another clinical study trial involving medical research or have participated within the last 30 days in a clinical study involving an investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more Treatment Emergent Adverse Event(s) (TEAEs) and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to 42 weeks
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Percent change from baseline in body weight | Baseline, Week 42
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve (AUC) of LY3841136 | Predose up to 42 weeks
Pharmacokinetics (PK): Maximum plasma concentration (Cmax) of LY3841136 | Predose up to 42 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/471555